CLINICAL TRIAL: NCT02262741
Title: A Phase I Study to Evaluate the Safety, Tolerability, and Efficacy of MEDI4736 in Combination With Tremelimumab in Subjects With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: A Phase I Study to Evaluate the Safety, Tolerability and Efficacy of MEDI4736 (Durvalumab) With Tremelimumab in Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4190C00011
Record Dates: First submitted 2014-10-02; First posted 2014-10-13 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MEDI4736 + tremelimumab (Experimental)
  Interventions: Biological: MEDI4736; Biological: tremelimumab

INTERVENTIONS:
Biological: MEDI4736 — MEDI4736 will be administered by IV infusion in combination with tremelimumab.
Biological: tremelimumab — Tremelimumab will be administered by IV infusion in combination with MEDI4736.

SUMMARY:
This is a multicenter, open-label, dose-exploration and dose-expansion study to evaluate the safety, tolerability, antitumor activity, PK, pharmacodynamics, and immunogenicity of MEDI4736 in combination with tremelimumab in subjects with recurrent/metastatic squamous cell carcinoma of the head and neck.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects
2. 18 years and older
3. Histologically or cytologically confirmed recurrent or metastatic squamous cell carcinoma of the head and neck (oral cavity, oropharynx, hypopharynx or larynx) that is incurable by local therapy.
4. Subjects who are treatment-naive or pretreated (prior anti-PD-1 or anti-PD-L1 required) in the recurrent/metastatic setting.
5. Subject eligibility will be based on PD-L1 expression as determined by a specified IHC assay.

Exclusion Criteria:

1. Any concurrent chemotherapy, immunotherapy, biologic, or hormonal therapy for cancer treatment, receipt of last dose of an approved anticancer therapy within 21 days
2. Concurrent or prior use of immunosuppressive medication within 14 days
3. Active or prior documented autoimmune or inflammatory disease within 3 years with some exceptions.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
Number of subjects reporting adverse events | Screening through 3 months after the last dose of study medication
Number of subjects reporting serious adverse events | Screening through 3 months after the last dose of study medication
Number of subjects experiencing dose-limiting toxicities | First dose of study medications through 4 weeks after the first dose of study medication
Change from Baseline in laboratory evaluations | Screening through 3 months after the last dose of study medication
Change from Baseline in electrocardiograms | Screening through 3 months through last dose of study medication
Change from Baseline in vital signs | Screening through 3 months after the last dose of study medication

SECONDARY OUTCOMES:
Objective Response Rate | Screening through 5 years after the last subject receives the first dose of study medication
Individual MEDI4736 concentrations | First dose of MEDI4736 through 3 months after the last dose of study medication
Number of subjects that develop changes in detectable antidrug antibodies to MEDI4736 | First dose of MEDI4736 through 6 months after the last dose of study medication
Disease Control Rate | Screening through 5 years after the last subject receives the first dose of study medication
Duration of Response | Screening through 5 years after the last subject receives the first dose of study medication
Progression Free Survival | Screening through 5 years after the last subject receives the first dose of study medication
Overall Survival | Screening through 5 years after the last subject receives the first dose of study medication
Individual tremelimumab concentrations | First dose of tremelimumab through 3 months after the last dose of study medication
MEDI4736 area under the concentration-curve | First dose of MEDI4736 through 3 months after the last dose of study medication
Tremelimumab area under the concentration-curve | First dose of tremelimumb through 3 months after the last dose of study medication
Number of subjects that develop changes in detectable antidrug antibodies to tremelimumab | First dose of tremelimumab through 6 months after the last dose of study medication

OTHER OUTCOMES:
Changes in Biomarkers | Screening through 3 months after the last patient receives the first dose of study medication
  Evaluate biomarkers that may correlate with clinical activity of MEDI4736 monotherapy and in combination with tremelimumab
Change from Baseline in Patient-Reported Outcomes | Screening through 5 years after the last patient receives the first dose of study medication

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (21):
- United States (19):
  - Research Site, Scottsdale, Arizona
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Aurora, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Orlando, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Fairway, Kansas
  - Research Site, New Orleans, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, New York, New York
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, San Antonio, Texas
  - Research Site, Fairfax, Virginia
- Canada (2):
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario

REFERENCES:
- [Derived] Algazi A, Papadopoulos KP, Tsai F, Hansen AR, Angra N, Das M, Sheth S, Siu LL. Safety and clinical activity of durvalumab combined with tremelimumab in recurrent/metastatic head and neck squamous cell carcinoma: a multicenter phase I study. ESMO Open. 2024 Aug;9(8):103646. doi: 10.1016/j.esmoop.2024.103646. Epub 2024 Jul 23. PMID 39043009